CLINICAL TRIAL: NCT01697124
Title: The Children in Action Feasibility Study
Acronym: CIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Theresa A Nicklas, Professor of Pediatrics, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H-20952; R21HD054836-02 (NIH)
Record Dates: First submitted 2012-09-17; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Obesity; Motor Activity
Keywords: Physical activity; children; Head Start; SPARK-EC
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SPARK-EC (Experimental): SPARK-EC curriculum for preschoolers offered instruction and practice in a comprehensive program designed to promote motor development through increased physical activity.
  Interventions: Behavioral: SPARK-EC

INTERVENTIONS:
Behavioral: SPARK-EC — The CIA study was a 5 month physical activity change intervention that utilized the SPARK-EC curriculum as the intervention. The SPARK-EC curriculum was designed to be a quality, comprehensive physical activity program for the preschool setting. Pre-and Post-intervention assessments were conducted

SUMMARY:
The Children in Action (CIA) program was a five month physical activity intervention. This intervention was a feasibility study with 3- to 5-year-olds enrolled in four Head Start centers. After baseline assessment, centers were matched by ethnicity and for number of participants and randomly assigned to either the intervention or the control condition. A total of 224 preschool children were randomly selected across the four centers. To evaluate the efficacy of the CIA intervention, the change in physical activity, gross motor skills and weight during the awake time and used mixed effect time-series regression models was compared. Observations did not show a statistical difference between intervention and control groups in physical activity level during the awake time, gross motor development or weight status. It was demonstrated that it is feasible to conduct the SPARK-EC curriculum among preschool children attending Head Start Centers but that an increased dose and/or longer intervention duration will be required to impact gross motor skills, weight status and physical activity levels during this critical early childhood development stage.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 years old
* attends Head Start
* African-American
* Hispanic-American

Exclusion Criteria:

* older than 5 years old
* does not attend Head Start
* race/ethnicity other than African-American or Hispanic-American
* has a disability or handicap that would prevent them from participating in physical activities

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 274 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical activity at post-intervention. | 8 months
  Mini-Mitter Actical, an accelerometer-based activity monitor, was used to assess physical activity of the preschool children. Unit of measurement was mean percentage of time spent in sedentary, light and moderate-vigorous physical activity each day.

SECONDARY OUTCOMES:
Change from baseline in gross motor skills at post intervention. | 8 months
  Gross motor skills were measured using the Test of Gross Motor Development. Unit of measurement was the Total Gross Motor Development percentile rank.
Body Mass Index | 8 months
  Body Mass Index was calculated using height and weight measures collected on the preschool children. Unit of measurement was kilograms (wt.)/meters squared (ht.).

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Nicklas, DrPH, Principal Investigator — Baylor College of Medicine